CLINICAL TRIAL: NCT02897362
Title: Sleep Dysfunction and Neurocognitive Outcomes in Adolescent ADHD
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00072033; 1K23MH108704-01A1 (NIH)
Record Dates: First submitted 2016-09-02; First posted 2016-09-13 (Estimated); Last update posted 2021-07-14 (Actual); Status verified 2021-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Sleep; Adolescents; Neurocognition; Polysomnography
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Adolescents with ADHD: Adolescents, male or female, ages 13-17, confirmed diagnosis of Attention Deficit Hyperactivity Disorder (inattentive, hyperactive/impulsive, or combined presentations), medically healthy, no comorbid psychiatric diagnosis other than ODD, intelligence within normal limits. Participants will complete 3 nights of ambulatory polysomnography at home and a neuropsychological assessment in the lab.
- Healthy Control Adolescents: Adolescents, male or female, ages 13-17, medically healthy, no psychiatric diagnoses, intelligence within normal limits. Participants will complete 3 nights of ambulatory polysomnography at home and a neuropsychological assessment in the lab.

SUMMARY:
This study seeks to characterize sleep physiology in adolescents with and without Attention deficit hyperactivity disorder (ADHD) and its relationship to differential neurocognitive and clinical outcomes within these groups.

DETAILED DESCRIPTION:
This project will involve recruitment of 30 adolescents with ADHD and a control group of 30 healthy adolescents without psychiatric diagnoses. Participants will participate in 3 phases: Screening visit, Washout/In-Home Sleep Study, and Neurocognitive Assessment visit. To ensure consistency in sleep schedules, the three nights of the sleep study will occur on weeknights during the school year. The neurocognitive assessment will occur during the afternoon following the final night of sleep assessment.

The 2-hour screening visit will be conducted at the Duke ADHD Clinic at 2608 Erwin Road, Pavilion East, Suite 300, Durham, NC 27705. During the screening visit, participants will undergo screening to evaluate eligibility for the study.

Eligible participants will enter the 48-hour Washout from stimulant medication (if applicable) and/or a 7-day washout from melatonin (if applicable). Following this washout, subjects will enter a 3-night Sleep Study Phase (At Home). Subjects not taking stimulant medication or melatonin will initiate 3 consecutive nights of ambulatory (in-home) PSG recording, beginning on the a Monday evening within 4 weeks of the screening visit. Subjects will be instructed to maintain usual sleep routines/behaviors for all study nights. In addition, subjects will be asked to complete a "sleep diary" each morning.

If subject is currently taking stimulant medication, they will be instructed to initiate a 48-hour washout period. If subject is currently taking melatonin, they will be instructed to initiate a 7-day washout period. Subjects will be instructed to discuss this option with their prescribing physician prior to initiating the study.

Subjects will be asked to return for a three hour neurocognitive assessment on the afternoon directly following the final night of the sleep study. In order to reduce interference with school attendance, this visit will be scheduled in the afternoon. Subjects will take breaks throughout the assessment.

Subjects will restart their ADHD medications on the morning following the neurocognitive assessment (if applicable).

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Between the ages of 13-17 years, inclusive;
* Free from significant medical/psychiatric conditions
* Cognitive functioning > 80 as assessed by the KBIT-II
* Willingness to comply with all study requirements; and
* Ability of child and parent/guardian to communicate verbally and in written form in English.

Inclusion for the ADHD group only:

* Confirmed diagnosis of ADHD, any subtype as determined by the MINI-KID
* Willingness to delay/suspend medication use for the 4-day duration of the study and 2 days prior to the sleep study phase.

Exclusion Criteria:

* History of chronic/significant medical condition
* Use of prescription medications for ADHD during the 2-day washout and/or 4-day study
* Current prescribed use of any other psychotropics, including non-stimulant medications for ADHD
* Current substance abuse or dependence or history within the last 6 months
* Estimated IQ < 80 as assessed by the KBIT-II
* First degree relative with psychosis or bipolar disorder;
* Parent/Guardian or child unable to communicate verbally and in written form in English; and
* Unable to comply with study requirements or otherwise unsuitable for participation in the opinion of the principal investigator

Exclusion for the ADHD group only:

* Meets criteria for any other Axis I Disorder (determined by the MINI-KID) besides ADHD or Oppositional Defiant Disorder (ODD)

Exclusion for the HEALTHY CONTROL group only:

* Meets criteria for any Axis I Disorder

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Adolescents with ADHD and healthy control adolescents
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2016-08; Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Objective sleep assessment | 3 consecutive nights
  Ambulatory polysomnographic measures of total sleep time, sleep onset latency, wake after sleep onset, and EEG spectral dynamics.

SECONDARY OUTCOMES:
Neurocognitive assessment | 1 day
  Computerized measure of neurocognition.
Executive functioning as measured by neurocognitive assessment | 1 day
  Measure of executive function

CONTACTS AND LOCATIONS:
Overall Officials: Jessica R Lunsford-Avery, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Child and Family Study Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lunsford-Avery JR, Carskadon MA, Kollins SH, Krystal AD. Sleep Physiology and Neurocognition Among Adolescents With Attention-Deficit/Hyperactivity Disorder. J Am Acad Child Adolesc Psychiatry. 2025 Feb;64(2):276-289. doi: 10.1016/j.jaac.2024.03.005. Epub 2024 Mar 12. PMID 38484795